CLINICAL TRIAL: NCT04719780
Title: A Randomized Controlled Trial of an Attachment Based Approach for Anxiety and Depression, Emotionally Focused Individual Therapy
Brief Title: An Attachment Based Approach for Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Paul University (Other)
Collaborators: International Centre for Excellence in Emotionally Focused Therapy (Unknown)
Responsible Party: Principal Investigator, Stephanie Wiebe, Assistant Professor, Saint Paul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1360.9/19
Record Dates: First submitted 2020-05-10; First posted 2021-01-22 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Depression, Anxiety
Keywords: Randomized control trial; Emotionally focused therapy; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Emotion-Focused Therapy

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled trial (RCT) carried out across three study sites (Ottawa, Denver, Victoria). We will have two study groups, treatment (n=44) and wait-list control (n=44). The wait-list control will be given an online transdiagnostic cognitive-behavioural treatment for depression and anxiety that has been empirically validated. The treatment condition group will be provided 12-15 sessions of Emotionally Focused Therapy for Individuals. Approximately 22 experienced EFT therapists will be given training in EFIT and will provide treatment to 2-3 clients each. Therapy will be carried out in person and/or online.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control Group (CBT) (Active Comparator): Individuals in this arm (n=44) are provided with a transdiagnostic cognitive-behavioural treatment for depression and anxiety (MoodGym) that has been empirically validated after their 15-week wait period is complete.
  Interventions: Behavioral: Self-Help CBT Training
- EFIT Group (Experimental): Individuals in the EFIT Group (n=44) will receive 12-15 sessions of EFIT in order to treat their symptoms of depression and anxiety.
  Interventions: Behavioral: Emotionally Focused Therapy for Individuals

INTERVENTIONS:
Behavioral: Emotionally Focused Therapy for Individuals — Emotionally Focused Therapy for Individuals (EFIT) is formulated as a transdiagnostic treatment to treat depression and anxiety, adapted from the well-studied Emotionally Focused Therapy. EFIT has been formulated as an attachment-based alternative to current cognitive approaches (e.g., Cognitive Behavioural Therapy). The strong evidence for insecure attachment as an underlying factor in psychopathology, especially depression and anxiety, positions this theory well as a foundational principle to support psychotherapy for these conditions.
  Arms: EFIT Group
Behavioral: Self-Help CBT Training — Individuals in the Waitlist Control Group will receive access to MoodGym, a self-help online program that helps teach CBT interventions. This access will last 15 weeks and is self-driven, meaning participants proceed through the program at their own pace.
  Other Names: MoodGym
  Arms: Waitlist Control Group (CBT)

SUMMARY:
The purpose of the current study is to examine the efficacy of Emotionally Focused Therapy for Individuals (EFIT) as a treatment for depression and anxiety. It is formulated as a trans-diagnostic treatment in line with the call for more transdiagnostic approaches to treat depression and anxiety given the many similarities in the underlying psychological and emotional factors of these disorders, the high levels of co-morbidity, and the preliminary success of transdiagnostic treatment approaches. EFIT has been formulated as an attachment-based alternative to current cognitive transdiagnostic approaches. The strong evidence for insecure attachment as an underlying factor in psychopathology, especially depression and anxiety, positions this theory well as a foundational principle to support psychotherapy for these conditions. EFIT has been formulated for the first time this year in the book that will serve as the therapy manual for this study. The current study aims to examine EFIT outcomes as compared to a control group (a wait-list control followed by online CBT intervention after the wait period). In particular, this research project aims to distinguish differences in initial and follow-up outcomes between EFIT versus control, and demonstrate significant changes in attachment/emotions and mechanisms of change across EFIT sessions. The primary hypotheses are outlined below.

DETAILED DESCRIPTION:
PROCEDURES

Recruitment Participants are recruited from the general population of individuals self-identifying as having symptoms of depression and/or anxiety in each study site (Ottawa, Denver, Victoria). Study advertisements are posted and circulated through post-secondary institutions, online, and within psychotherapy treatment centres. Participants experiencing depression and/or anxiety are invited to contact the research coordinator of the project via the email listed on recruitment material. All interested participants receive a telephone screen by research research assistants to assess potential eligibility. Participants who are deemed potentially eligible are informed that they will be contacted by an assessor to be invited for an initial study assessment session to determine final eligibility.

Baseline assessment Assessors are individuals with clinical experience in psychotherapy or counselling at each of the study sites. Informed consent is reviewed and participants have the opportunity to have all their questions and concerns addressed. Assessors administer the diagnostic criteria modules of the ADIS-5 during this session. Assessments take place either within the private practice locations at each study site or the university offices of the investigators in a research session lasting approximately 1-2 hours. During the pandemic while it is not safe to meet in person, secure encrypted video call platforms are used to hold these sessions. Responses are evaluated by the assessors' supervisors, at which point final eligibility is determined. The assessments and therapy take place either within the private practice locations at each study site as specified or the university offices of the co-investigators, or online using a secure encrypted video call platform when it is unsafe to meet for in-person sessions due to the pandemic. After completion of the baseline assessment session, eligible participants are given access to an online questionnaire to complete at their own convenience. After completion of the questionnaire, participants are randomly assigned to study condition.

Random assignment Once participants have been deemed eligible to take part, and have completed the baseline questionnaire, they are randomly assigned to the EFIT (treatment) condition or the waitlist plus online CBT (control group) condition by the research co-ordinator. A list of numbers (i.e., 1-40 for Ottawa, 1-28 for Victoria, and 1-20 for Denver) are generated for each city, reflecting the total number of EFIT and control clients for that city. Within those groups, a separate randomized list (i.e., 20 total numerical values for Ottawa, 14 for Victoria, and 10 for Denver) is generated using Research Randomizer, an online tool for random assignment that has been used in previous RCT studies. As participants are deemed eligible, they are added onto the list and their number will determine whether they will take part in either the EFIT intervention or the control group.

Interventions:

EFIT Treatment Group Twenty-two experienced EFT therapists trained in the EFIT model will provide 15 sessions of EFIT treatment to approximately 2 clients each. Therapy will be carried out in private practices or the university offices of researchers located in each of the study sites, or online using a secure encrypted video call platform when not possible to meet in person due to the pandemic. Each site is associated with an EFT centre: Ottawa Institute of Couple and Family Therapy in Ottawa, Centre for EFT Vancouver Island in Victoria, and Colorado Centre for EFT in Denver. Study therapists will receive an average of 1 hour of supervision per week in groups of 3-4 therapists. Each therapy session will be video recorded and treatment fidelity will be confirmed through the coding of video tapes. After each therapy session, therapists will ask participants to complete a brief online questionnaire that takes approximately 10 minutes to complete. The link to the online questionnaire will be sent to each therapist by the research co-ordinator.

Wait-List plus online CBT Control Group Participants randomly assigned to the wait-list control group will wait 15 weeks, following which time they will be given an online transdiagnostic cognitive-behavioural treatment (MoodGym) for depression and anxiety that has been empirically validated after they have completed the 15-week wait period. They will be given access to complete 15 weeks of the online intervention. These participants will also be requested to complete a brief online questionnaire on a weekly basis - this questionnaire is identical to the questionnaire given to EFIT participants after each therapy session with the exception that it does not include the Working Alliance Inventory (WAI) or the Post-session Resolution Questionnaire (PSRQ) as these questionnaires are only relevant to therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder with co-morbid symptoms of anxiety
* Inclusion cut offs: Participants must score in the mild-to severe range on BDI-II and mild-moderate on the BAI
* At least 18 years old

Exclusion Criteria:

* Psychotropic medication change in 6 weeks prior to enrollment or anticipated during the study period (this allows us to include people who are taking a medication but mitigates the risk of medication changes as a problematic factor; assessed in phone screen)
* Current DSM diagnosis of bipolar disorder, schizophrenia-spectrum disorder, PTSD, eating disorder, personality disorder, or substance abuse or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5) | Change from baseline to completion of the 15 week intervention.
  The ADIS-5 is a structured interview intended to help clinicians diagnose psychological disorders based on DSM-5 criteria. The ADIS-5 also allows for differential diagnosis and has been widely used in clinical research. Assessors will administer the ADIS-5 and determine whether or not the participants the criteria for a diagnosis of anxiety and/or depression, and to assess change upon completion of the 15-week intervention.
Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5) | Change from baseline to completion of the 15 week wait period.
  The ADIS-5 is a structured interview intended to help clinicians diagnose psychological disorders based on DSM-5 criteria. The ADIS-5 also allows for differential diagnosis and has been widely used in clinical research. Assessors will administer the ADIS-5 and determine whether or not the participants the criteria for a diagnosis of anxiety and/or depression, and to assess change at post 15-week wait period.
Beck Depression Inventory-2 (BDI-2) | Change from baseline to week 5, week 7, completion of 15-week wait period (control condition), and 3, 6, 9 and 12 months following completion of the wait-period.
  The Beck Depression Inventory-2 is a 21-item self-report questionnaire used to assess the severity of depressive symptoms (e.g., sadness, guilt, crying, suicidal thoughts, etc.). Participants are presented with a list of themes and are asked to choose a statement that best fits their mood over the past two weeks. Each statement has a corresponding numerical value. The sum all statements are calculated for scoring purposes. A score of 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression, and a score above 29 indicates severe depression. Participants will complete this questionnaire in paper format at the baseline and post assessment sessions. EFIT participants will also complete the BDI after session 5 and 7.
Beck Depression Inventory-2 (BDI-2) | Change from baseline to week 5, week 7, completion of 15-week intervention, and 3, 6, 9 and 12 months following the intervention.
  The Beck Depression Inventory-2 is a 21-item self-report questionnaire used to assess the severity of depressive symptoms (e.g., sadness, guilt, crying, suicidal thoughts, etc.). Participants are presented with a list of themes and are asked to choose a statement that best fits their mood over the past two weeks. Each statement has a corresponding numerical value. The sum all statements are calculated for scoring purposes. A score of 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression, and a score above 29 indicates severe depression. Participants will complete this questionnaire in paper format at the baseline and post assessment sessions. EFIT participants will also complete the BDI after session 5 and 7.
Beck Anxiety Inventory (BAI) | Change from baseline to week 5, week 7, and completion of 15-week wait period (control condition) and at 3, 6, 9, and 12 months after completing the wait-period
  The Beck Anxiety Inventory is a 21-item self-report questionnaire used to assess common symptoms of anxiety (e.g., rapid heartbeat, sweating, numbness, trembling, etc.). Participants are presented with a list of common symptoms of anxiety and are asked to note how much they experienced each over the past week from a four item Likert scale ("not at all", "mildly", "moderately", and "severely"). The total score is calculated by finding the sum of all 21 items; a score of 0-21 indicated low anxiety, 22-35 indicates moderate anxiety, and a score of 36 and above indicates potentially concerning levels of anxiety. Both of the Beck inventories used in this study have been widely used in clinical research and possess good reliability and validity. Participants will complete this questionnaire in paper format at the baseline and post assessment sessions. EFIT participants will also complete the BDI-2 after session 5 and 7.
Beck Anxiety Inventory (BAI) | Change from baseline to week 5, week 7 and completion of 15-week intervention, and at 3, 6, 9, and 12 months after completing the intervention
  The Beck Anxiety Inventory is a 21-item self-report questionnaire used to assess common symptoms of anxiety (e.g., rapid heartbeat, sweating, numbness, trembling, etc.). Participants are presented with a list of common symptoms of anxiety and are asked to note how much they experienced each over the past week from a four item Likert scale ("not at all", "mildly", "moderately", and "severely"). The total score is calculated by finding the sum of all 21 items; a score of 0-21 indicated low anxiety, 22-35 indicates moderate anxiety, and a score of 36 and above indicates potentially concerning levels of anxiety. Both of the Beck inventories used in this study have been widely used in clinical research and possess good reliability and validity. Participants will complete this questionnaire in paper format at the baseline and post assessment sessions. EFIT participants will also complete the BDI-2 after session 5 and 7.
Outcome Questionnaire-30.2 | Change from baseline, to across each weekly treatment session for 15 weeks, to after completion of the 15-week intervention, and at 3, 6, 9, and 12 months after completing the intervention
  The Outcome Questionnaire-30.2 is a brief 30-item instrument intended to measure client progress before, during, and following clinical interventions. This questionnaire is was adapted from the OQ-45, is highly sensitive to session-by-session changes, and possesses high levels of reliability and validity. Over the course of the study, this questionnaire will be repeatedly administered in order to monitor participants' progress through the EFIT and waitlist conditions. This questionnaire will also be administered during the 4 follow-up time points.
Outcome Questionnaire-30.2 | Change from baseline, to across each week for 15 weeks, to after completion of the 15-week wait-period, and at 3, 6, 9, and 12 months after completing the 15-week wait-period.
  The Outcome Questionnaire-30.2 is a brief 30-item instrument intended to measure client progress before, during, and following clinical interventions. This questionnaire is was adapted from the OQ-45, is highly sensitive to session-by-session changes, and possesses high levels of reliability and validity. Over the course of the study, this questionnaire will be repeatedly administered in order to monitor participants' progress through the EFIT and waitlist conditions. This questionnaire will also be administered during the 4 follow-up time points.
Patient-Reported Outcomes Measurement Information System-Anxiety Scale (PROMIS Anxiety) | Change from baseline, to across each weekly treatment session for 15 weeks, to after completion of the 15-week intervention, and at 3, 6, 9, and 12 months after completing the intervention
  The Patient-Reported Outcomes Measurement Information System-Anxiety scale is an 8-item tool designed to measure participants' self-reported anxiety symptoms over the past week. Participants are asked to respond to eight anxiety-related statements on a 5-point Likert scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=always).
Patient-Reported Outcomes Measurement Information System-Anxiety Scale (PROMIS Anxiety) | Change from baseline, to across each week for 15 weeks, to after completion of the 15-week wait-period, and at 3, 6, 9, and 12 months after completing the 15-week wait-period.
  The Patient-Reported Outcomes Measurement Information System-Anxiety scale is an 8-item tool designed to measure participants' self-reported anxiety symptoms over the past week. Participants are asked to respond to eight anxiety-related statements on a 5-point Likert scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=always).
Patient-Reported Outcomes Measurement Information System-Depression Scale (PROMIS Depression) | Change from baseline, to across each weekly treatment session for 15 weeks, to after completion of the 15-week intervention, and at 3, 6, 9, and 12 months after completing the intervention
  The Patient-Reported Outcomes Measurement Information System-Depression scale is an 8-item scale used to measure participants' self-reported depression symptoms over the past week. Participants are asked to respond to eight depression-related statements on the same 5-point Likert scale as the PROMIS-Anxiety measure.
Patient-Reported Outcomes Measurement Information System-Depression Scale (PROMIS Depression) | Change from baseline, to across each week for 15 weeks, to after completion of the 15-week wait-period, and at 3, 6, 9, and 12 months after completing the 15-week wait-period.
  The Patient-Reported Outcomes Measurement Information System-Depression scale is an 8-item scale used to measure participants' self-reported depression symptoms over the past week. Participants are asked to respond to eight depression-related statements on the same 5-point Likert scale as the PROMIS-Anxiety measure.

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire-Short Form | Baseline
  It is a 28-item self-report scale that measures self-reported occurrence of maltreatment in childhood and adolescence. Participants will be asked to answer statements with a corresponding Likert scale value. A total of five factors are included in this measure: sexual abuse, physical abuse, emotional abuse, emotional neglect, and physical neglect; each factor has its own cut-off score.
Trauma Symptom Inventory-2 | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The TSI-2 evaluates post-traumatic stress symptomatology and other long-term effects of trauma (e.g., dissociation, insecure attachment styles, somatization, etc.) on a 4-point Likert Scale. Participants are asked to rate 136 brief statements based on their level of agreement.
Trauma Symptom Inventory-2 | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The TSI-2 evaluates post-traumatic stress symptomatology and other long-term effects of trauma (e.g., dissociation, insecure attachment styles, somatization, etc.) on a 4-point Likert Scale. Participants are asked to rate 136 brief statements based on their level of agreement.
Experiences in Close Relationships Questionnaire (ECR) | Change from baseline, to across each weekly treatment session for 15 weeks, to after completion of the 15-week intervention, and at 3, 6, 9, and 12 months after completing the intervention
  The Experiences in Close Relationships Questionnaire is a 12 item questionnaire that measures individuals' attachment to romantic partners; the current study, however, received special permission to revise the wording and change "romantic partner" to "loved one". The ECR contains two scales, each containing 18 items: attachment anxiety, and attachment avoidance. The questionnaire is scored on a 7-point scale (1=strongly disagree, 7=strongly agree).
Experiences in Close Relationships Questionnaire (ECR) | Change from baseline, to across each week for 15 weeks, to after completion of the 15-week wait-period, and at 3, 6, 9, and 12 months after completing the 15-week wait-period.
  The Experiences in Close Relationships Questionnaire is a 12 item questionnaire that measures individuals' attachment to romantic partners; the current study, however, received special permission to revise the wording and change "romantic partner" to "loved one". The ECR contains two scales, each containing 18 items: attachment anxiety, and attachment avoidance. The questionnaire is scored on a 7-point scale (1=strongly disagree, 7=strongly agree).
Reflective Function Questionnaire-8 (RFQ) | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Reflective Function Questionnaire-8 is the short form version of the longer 54-item measure. This questionnaire is used to measure the degree of certainty the participants experience regarding their awareness of their own and others' mental states. Questions on the RFQ are measured on a 7-point Likert scale (1=strongly disagree, 7=strongly agree).
Reflective Function Questionnaire-8 (RFQ) | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Reflective Function Questionnaire-8 is the short form version of the longer 54-item measure. This questionnaire is used to measure the degree of certainty the participants experience regarding their awareness of their own and others' mental states. Questions on the RFQ are measured on a 7-point Likert scale (1=strongly disagree, 7=strongly agree).
Inventory of Interpersonal Problems-32 | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Inventory of Interpersonal Problems-32 is a self-report questionnaire that identifies participants' sources of interpersonal distress generally.. The IIP-32 is a short form of the original 64-item measure. For the first 20 items, participants are asked to rate their level of difficulty with diverse situations on a 5-point Likert scale (0=not at all, 5=extremely). For the remaining items, participants are asked to rate "things [they] do too much" (e.g., please others) on a similar scale. The IIP has been used in psychotherapy sessions wherein clients and therapists complete the measure in order to focus on specific interpersonal difficulties experienced by the client.
Inventory of Interpersonal Problems-32 | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Inventory of Interpersonal Problems-32 is a self-report questionnaire that identifies participants' sources of interpersonal distress generally.. The IIP-32 is a short form of the original 64-item measure. For the first 20 items, participants are asked to rate their level of difficulty with diverse situations on a 5-point Likert scale (0=not at all, 5=extremely). For the remaining items, participants are asked to rate "things [they] do too much" (e.g., please others) on a similar scale. The IIP has been used in psychotherapy sessions wherein clients and therapists complete the measure in order to focus on specific interpersonal difficulties experienced by the client.
Difficulties in Emotion Regulation Scale | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Difficulties in Emotion Regulation Scale is a 32-item questionnaire used to measure participants' difficulties with emotion regulation. The DERS contains six subscales: non-acceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Participants are asked to indicate how often the 32 presented statements apply to them. Items are scored on a 5-point Likert scale (1=almost never 0-10%, 5=almost always 91-100%).
Difficulties in Emotion Regulation Scale | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Difficulties in Emotion Regulation Scale is a 32-item questionnaire used to measure participants' difficulties with emotion regulation. The DERS contains six subscales: non-acceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Participants are asked to indicate how often the 32 presented statements apply to them. Items are scored on a 5-point Likert scale (1=almost never 0-10%, 5=almost always 91-100%).
Leuven Affect and Pleasure Scale | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Leuven Affect and Pleasure Scale instrument asks participants to indicate the extent to which they experienced 16 feelings and emotionally-saturated situations (e.g., looking forward to something). Participants are provided with a 10-point Likert scale (0=not at all, 10=very much).
Leuven Affect and Pleasure Scale | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Leuven Affect and Pleasure Scale instrument asks participants to indicate the extent to which they experienced 16 feelings and emotionally-saturated situations (e.g., looking forward to something). Participants are provided with a 10-point Likert scale (0=not at all, 10=very much).
Rosenberg Self-Esteem Scale | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Rosenberg Self-Esteem Scale is a 10-item instrument that is used to measure positive and negative feelings relating to self-worth. Items are scored on a 4-point Likert scale (1=strongly agree, 4=strongly disagree). In order to score responses, researchers are advised to reverse score items 2, 5, 6, 8, and 9 before summing participants' total scores. Higher scores on the scale indicate higher levels of self-esteem.
Rosenberg Self-Esteem Scale | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Rosenberg Self-Esteem Scale is a 10-item instrument that is used to measure positive and negative feelings relating to self-worth. Items are scored on a 4-point Likert scale (1=strongly agree, 4=strongly disagree). In order to score responses, researchers are advised to reverse score items 2, 5, 6, 8, and 9 before summing participants' total scores. Higher scores on the scale indicate higher levels of self-esteem.
Patient-Reported Outcomes Measurement Information System-Meaning (PROMIS Meaning) | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Patient-Reported Outcomes Measurement Information System-Meaning instrument is an 8-item questionnaire intended to evaluate individuals' sense of purpose and meaning in life. Participants are asked to rate their level of agreement with eight statements based on a 5-point Likert scale (1=strongly disagree, 5=strongly agree).
Patient-Reported Outcomes Measurement Information System-Meaning (PROMIS Meaning) | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Patient-Reported Outcomes Measurement Information System-Meaning instrument is an 8-item questionnaire intended to evaluate individuals' sense of purpose and meaning in life. Participants are asked to rate their level of agreement with eight statements based on a 5-point Likert scale (1=strongly disagree, 5=strongly agree).
Multi-dimensional Assessment of Interoceptive Awareness | Change from baseline to week 5 and week 7, and completion of 15-week wait period (control condition) and across to 3, 6, 9, and 12 month follow-up time points
  The Multi-dimensional Assessment of Interoceptive Awareness is a 37-item questionnaire that assesses interoceptive body awareness, a key element of emotion regulation. The measure consists of 8 subscales: Noticing, Not-distracting, Not-worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening and Trusting. Higher scores indicate better interoceptive awareness aspects of affect regulation.
Multi-dimensional Assessment of Interoceptive Awareness | Change from baseline to week 5, week 7, and completion of 15-week intervention, and across 3, 6, 9, and 12 month follow-up time points
  The Multi-dimensional Assessment of Interoceptive Awareness is a 37-item questionnaire that assesses interoceptive body awareness, a key element of emotion regulation. The measure consists of 8 subscales: Noticing, Not-distracting, Not-worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening and Trusting. Higher scores indicate better interoceptive awareness aspects of affect regulation.
Post Session Resolution Questionnaire (PSQR) | Weekly for 15 weeks of the experimental condition
  The Post Session Resolution Questionnaire is a measurement tool intended to evaluate the fit of session topics to participants' established therapeutic goals. The questionnaire also allows participants to rate how much they thought a clinical session allowed them to progress towards the resolution of their presenting concerns. Three our of the four items in the PSQR operate on a 5-point Likert scale, the fourth item uses a 7-point scale.
Working Alliance Inventory | Weekly for 15 weeks of the experimental condition
  The Working Alliance Inventory is 12-item clinical tool which measures three key features of the therapeutic alliance: 1) agreement on tasks for therapy, 2) agreement on therapeutic goals, and 3) the development of a strong therapeutic relationship. Participants are presented with a list of statements and are asked to rate the frequency with which these statements reflect the therapeutic alliance they share with their therapist. A 5-point Likert scale is used to rate the participants' perceptions of their therapeutic alliance.
Sociodemographic Questionnaire | Baseline
  This questionnaire collects participants' demographic information, such as age, gender, location, income, marital status, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wiebe, PhD, Principal Investigator — Saint Paul University
Locations (3):
- University of Colorado Denver, Denver, Colorado, United States
- Canada (2):
  - Vancouver Island Centre for Emotionally Focused Therapy, Nanaimo, British Columbia
  - Saint Paul University, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Demyttenaere K, Mortier P, Kiekens G, Bruffaerts R. Is there enough "interest in and pleasure in" the concept of depression? The development of the Leuven Affect and Pleasure Scale (LAPS). CNS Spectr. 2019 Apr;24(2):265-274. doi: 10.1017/S1092852917000578. Epub 2017 Nov 9. PMID 29117870
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Horowitz LM, Rosenberg SE, Baer BA, Ureno G, Villasenor VS. Inventory of interpersonal problems: psychometric properties and clinical applications. J Consult Clin Psychol. 1988 Dec;56(6):885-92. doi: 10.1037//0022-006x.56.6.885. No abstract available. PMID 3204198
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Derived] Wiebe SA, Johnson SM, Allan R, Campbell TL, Greenman PS, Fairweather DR, Ismail M, Tasca GA. A randomized controlled trial of emotionally focused individual therapy (EFIT) for depression and anxiety. Psychotherapy (Chic). 2025 Sep;62(3):414-423. doi: 10.1037/pst0000586. Epub 2025 Jul 10. PMID 40638305
- See also: Applied longitudinal data analysis: Modeling change and event occurrence — https://books.google.ca/books?hl=en&lr=&id=PpnA1M8VwR8C&oi=fnd&pg=PA1&dq=Singer,+J.+D.+%26+Willett,+J.+B.+(2003).+Applied+longitudinal+data+analysis:+Modeling+change+and+event+occurrence.+New+York,+NY:+Oxford.&ots=N5tbqA7DrN&sig=Lqm7fbD0tq4SVnCl2j1UoGJRPHc#v=onepage&q&f=false
- See also: Attachment Theory in Practice: Emotionally Focused Therapy with Individuals, Couples and Families — https://books.google.ca/books?hl=en&lr=&id=6Rx9DwAAQBAJ&oi=fnd&pg=PP1&dq=Johnson,+S.+M.+(2019).+Attachment+Theory+in+Practice:+Emotionally+Focused+Therapy+with+Individuals,+Couples+and+Families.+New+York,+Guilford+Press.&ots=fOp3nJzJmL&sig=Rm9FbERvsHwCVEN-jNTtmazSpWY&redir_esc=y#v=onepage&q=Johnson%2C%20S.%20M.%20(2019).%20Attachment%20Theory%20in%20Practice%3A%20Emotionally%20Focused%20Therapy%20with%20Individuals%2C%20Couples%20and%20Families.%20New%20York%2C%20Guilford%20Press.&f=false
- See also: Childhood Trauma Questionnaire: A retrospective self-report — https://www.scienceopen.com/document?vid=db039366-86cf-448f-850c-f62f824bae8c